CLINICAL TRIAL: NCT00265590
Title: Phenotype-Genotype Correlation in Aniridia
Brief Title: Correlation of Gene Abnormalities and Clinical Manifestations of Aniridia
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060044; 06-EI-0044
Record Dates: First submitted 2005-12-14; First posted 2005-12-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-03

CONDITIONS: Aniridia
Keywords: Aniridia; PAX6; Keratopathy; Limbal Stem Cell Deficiency; Molecular Genetics
MeSH Terms: conditions — Aniridia; Limbal Stem Cell Deficiency

SUMMARY:
This study will examine specific gene changes in patients with aniridia, a disease in which the iris (colored part of the eye) is absent or partially absent, and will correlate the changes with clinical manifestations of the disease. In aniridia, the eye often appears to have no color, but only a larger than normal pupil. Patients may have impaired vision and cataracts, glaucoma, nystagmus (rapid, involuntary eye movements), photophobia (light sensitivity), displaced lens, underdeveloped retina, and thickened cornea. This study will focus particularly on corneal changes.

Patients 4 years old and older with aniridia may be eligible for this study. Candidates are screened with a family history and complete eye examination, including the following:

* Visual acuity testing using a vision chart.
* Eye pressure measurement.
* Fundus photography to examine the back of the eye: The pupils are dilated and special photographs of the inside of the eye are taken to evaluate the retina and measure changes that may occur over time. The camera flashes a bright light into the eye for each picture.
* Slit lamp examination: Evaluation of the front part of the eye with a special microscope called a slit lamp biomicroscope.
* Corneal thickness measurement.

Participants have blood drawn for genetic testing related to aniridia. Relevant medical information, including disease severity and complications, is obtained over time. Family members may also be requested to provide blood samples for genetic testing.

DETAILED DESCRIPTION:
This project, Phenotype-Genotype Correlation in aniridia, will study the specific mutations in patients with aniridia and attempt to make a phenotype-genotype correlation. Specifically, the study will determine whether specific mutations are more prevalent in aniridic patients who have a predominant involvement of the corneal epithelium. A blood sample will be collected from each individual for isolation of DNA and the PAX6 gene will be sequenced and analyzed. The principal investigator is Brian Brooks and the associated investigators are James Fielding Hejtmancik at the OMGS/OGVFB/NEI and Chi-Chao Chan, LI/NEI. Associate Investigators at collaborating institutions include Edward Holland (University of Cincinnati) and Ali Djalilian (University of Illinois, Chicago).

ELIGIBILITY:
* Patients that meet diagnostic criteria for aniridia will be recruited from the NEI and Collaborating clinics. While diagnosis of aniridia is not expected to create significant difficulty, every attempt will be made to document the clinical status of each family member included in the study, and to document the clinical syndrome in at least one affected individual by slit lamp photography. A total of 100 subjects will be recruited for this study. There are no specific exclusion criteria other than young age (less than 4 years old) which may pose difficulty in obtaining blood.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-12-07; Study Completion 2008-10-03

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Background] Nelson LB, Spaeth GL, Nowinski TS, Margo CE, Jackson L. Aniridia. A review. Surv Ophthalmol. 1984 May-Jun;28(6):621-42. doi: 10.1016/0039-6257(84)90184-x. PMID 6330922
- [Background] Elsas FJ, Maumenee IH, Kenyon KR, Yoder F. Familial aniridia with preserved ocular function. Am J Ophthalmol. 1977 May;83(5):718-24. doi: 10.1016/0002-9394(77)90139-8. PMID 868970
- [Background] Mintz-Hittner HA, Ferrell RE, Lyons LA, Kretzer FL. Criteria to detect minimal expressivity within families with autosomal dominant aniridia. Am J Ophthalmol. 1992 Dec 15;114(6):700-7. doi: 10.1016/s0002-9394(14)74048-6. PMID 1463039